CLINICAL TRIAL: NCT07155109
Title: The Effects of Different Intraperitoneal Pressures on Optic Nerve Sheath Diameter in Laparoscopic Gyneco-oncologic Surgeries
Brief Title: Different Intraperitoneal Pressures on Optic Nerve Sheath Diameter in Laparoscopic Surgeries
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Zeynep Koc, principal investigator, Diskapi Yildirim Beyazit Education and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: ZeynepKoc005
Record Dates: First submitted 2025-08-27; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Intracranial Pressure Increase; Abdominal Pain; Head Pain
Keywords: Intracranial Pressure; optic nerve; laparascopy; gyneco-oncologic surgery; low pressure
MeSH Terms: conditions — Intracranial Hypertension; Abdominal Pain; Headache

STUDY DESIGN:
Intervention Model Description: In laparoscopic gyneco-oncological surgeries, one group will receive low intraperitoneal pressure, while the other group will receive standart intraperitoneal pressure.
Who Masked: Participant
Masking Description: The investigator will be blinded to whether low or intraperitoneal pressure is applied to the patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Pressure Group (Experimental): In laparoscopic gyneco-oncological surgeries, low pressure group received below 12 mmHg intraperitoneal pressure.
  Interventions: Other: Low pressure group
- Normal Pressure Group (Experimental): In laparoscopic gyneco-oncological surgeries, normal pressure group received 12 and abowe 12 mmHg intraperitoneal pressure.
  Interventions: Other: Normal pressure group

INTERVENTIONS:
Other: Low pressure group — In laparoscopic gyneco-oncological surgeries, low pressure group will receive below 12 mmHg intraperitoneal pressure.
  Arms: Low Pressure Group
Other: Normal pressure group — In laparoscopic gyneco-oncological surgeries, normal pressure group will receive 12 and abowe 12 mmHg intraperitoneal pressure.
  Arms: Normal Pressure Group

SUMMARY:
The aim of this study is to investigate the effects of low and normal intraperitoneal pressures on intraoperative optic nerve sheath diameter in laparoscopic gyneco-oncologic surgeries.

DETAILED DESCRIPTION:
Gynecological surgeries are minimally invasive procedures. The establishment of pneumoperitoneum, special patient positioning, and surgical stimulation can induce a stress response in patients. Carbon dioxide (CO₂) pneumoperitoneum and the Trendelenburg position lead to increases in intra-abdominal, intrathoracic, and airway pressures, which in turn may directly or indirectly cause elevations in intracranial and intraocular pressures.

During the perioperative period, the optic nerve sheath diameter (ONSD), measured ultrasonographically, is used as a reliable method to estimate intracranial pressure (ICP). Monitoring ICP under anesthesia may help prevent neurological complications such as neurological deterioration and optic neuropathy. Furthermore, studies have demonstrated ICP changes in robotic and laparoscopic gynecologic surgeries through ultrasonographic measurement of ONSD.

Traditionally, laparoscopic abdominal surgeries are performed using intraperitoneal pressures ranging between 10 and 18 mmHg. Lower intra-abdominal pressures have been associated with reduced postoperative pain, improved pulmonary parameters, and a decreased risk of gas embolism. However, the data on these outcomes remain limited.

In this study, we aimed to investigate the effect of pressures above and below 12 mmHg on the optic nerve sheath diameter-and consequently on intracranial pressure-in patients undergoing laparoscopic gynecologic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Laparoscopic gyneco-oncological surgeries
* Female patients aged 18-65 years
* ASA physical status classification I-II-III patients

Exclusion Criteria:

* Patients with diabetic retinopathy
* Patients with glaucoma
* Patients with cerebrovascular disease
* Pregnant women
* Patients with known allergy to anaesthetic agents
* Morbidly obese patients with BMI > 40

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The study will be conducted in gyneco-oncological surgeries. The patient group will consist exclusively of female patients.
Enrollment: 100 (Estimated)
Dates: Start 2025-08-30 (Estimated); Primary Completion 2025-10-10 (Estimated); Study Completion 2025-10-20 (Estimated)

PRIMARY OUTCOMES:
Measurement of optic nerve sheath diameter (ONSD) | 30 minutes after introducing pneumoperitoneum and position change
  ONSD will be measured in the supine position by ulrasonographic measurement.After obtaining optimal contrast between the retrobulbar echogenic fat tissue and the vertical hypoechoic band, the ONSD will be measured 3 mm behind the optic disc using an electronic caliper. The final ONSD value was calculated by averaging 4 measured values: measured values of transverse and sagittal plane of both eyes.

SECONDARY OUTCOMES:
Measurement of optic nerve sheath diameter (ONSD) | The baseline ONSD measurement will be performed 5 minutes after endotracheal intubation
  ONSD will be measured by ulrasonographic measurement.After obtaining optimal contrast between the retrobulbar echogenic fat tissue and the vertical hypoechoic band, the ONSD will be measured 3 mm behind the optic disc using an electronic caliper. The final ONSD value was calculated by averaging 4 measured values: measured values of transverse and sagittal plane of both eyes.
Measurement of optic nerve sheath diameter (ONSD) | 5 minutes after introducing pneumoperitoneum and position change
  ONSD will be measured in the supine position by ulrasonographic measurement.After obtaining optimal contrast between the retrobulbar echogenic fat tissue and the vertical hypoechoic band, the ONSD will be measured 3 mm behind the optic disc using an electronic caliper. The final ONSD value was calculated by averaging 4 measured values: measured values of transverse and sagittal plane of both eyes.
Measurement of optic nerve sheath diameter (ONSD) | 60 minutes after introducing pneumoperitoneum and position change
  ONSD will be measured by ulrasonographic measurement.After obtaining optimal contrast between the retrobulbar echogenic fat tissue and the vertical hypoechoic band, the ONSD will be measured 3 mm behind the optic disc using an electronic caliper. The final ONSD value was calculated by averaging 4 measured values: measured values of transverse and sagittal plane of both eyes.
Measurement of optic nerve sheath diameter (ONSD) | 90 minutes after introducing pneumoperitoneum and position change
  ONSD will be measured by ulrasonographic measurement.After obtaining optimal contrast between the retrobulbar echogenic fat tissue and the vertical hypoechoic band, the ONSD will be measured 3 mm behind the optic disc using an electronic caliper. The final ONSD value was calculated by averaging 4 measured values: measured values of transverse and sagittal plane of both eyes.
Measurement of optic nerve sheath diameter (ONSD) | The ONSD measurement will be performed 5 minutes after the pneumoperitoneum is released and the Trendelenburg position is corrected.
  ONSD will be measured in the supine position by ulrasonographic measurement.After obtaining optimal contrast between the retrobulbar echogenic fat tissue and the vertical hypoechoic band, the ONSD will be measured 3 mm behind the optic disc using an electronic caliper. The final ONSD value was calculated by averaging 4 measured values: measured values of transverse and sagittal plane of both eyes.

OTHER OUTCOMES:
numerical rating scale (NRS) at rest | popstoperative 1. hour
  Recording the patient's pain at rest on the Numerical Rating Scale (NRS) by asking the patient
numerical rating scale (NRS) at rest | popstoperative 8. hours
  Recording the patient's pain at rest on the Numerical Rating Scale (NRS) by asking the patient
postoperative nosia and vomiting (PONV) | popstoperative 1. hour
  Recording the presence or absence of nausea and vomiting in the patient within the first 24 hours postoperatively
postoperative nosia and vomiting (PONV) | popstoperative 8. hours
  Recording the presence or absence of nausea and vomiting in the patient within the first 24 hours postoperatively
headache | popstoperative 8. hours
  The presence or absence of headache will be assessed and documented.

CONTACTS AND LOCATIONS:
Locations (1):
- Zeynep Koç, Yenimahalle, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The optic nerve sheath diameter measurements will be shared with other researchers in the later stages of the study.

REFERENCES:
- [Background] Lee YY, Lee H, Park HS, Kim WJ, Baik HJ, Kim DY. Optic nerve sheath diameter changes during gynecologic surgery in the Trendelenburg position: comparison of propofol-based total intravenous anesthesia and sevoflurane anesthesia. Anesth Pain Med (Seoul). 2019 Oct 31;14(4):393-400. doi: 10.17085/apm.2019.14.4.393. PMID 33329767
- [Background] Geng W, Chen C, Sun X, Huang S. Effects of sevoflurane and propofol on the optic nerve sheath diameter in patients undergoing laparoscopic gynecological surgery: a randomized controlled clinical studies. BMC Anesthesiol. 2021 Jan 27;21(1):30. doi: 10.1186/s12871-021-01243-7. PMID 33504329
- [Background] Kim SH, Kim HJ, Jung KT. Position does not affect the optic nerve sheath diameter during laparoscopy. Korean J Anesthesiol. 2015 Aug;68(4):358-63. doi: 10.4097/kjae.2015.68.4.358. Epub 2015 Jul 28. PMID 26257848